CLINICAL TRIAL: NCT05807191
Title: The Effect of Using Clinical Guidelines on Kangaroo Care in Premature Infants on Newborn and Maternal Outcomes: A Randomized Controlled Trial
Brief Title: The Effect of Using Clinical Guidelines on Kangaroo Care on Newborn and Maternal Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SelcukU-12-2022
Record Dates: First submitted 2022-12-20; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Premature Infants
Keywords: Kangaroo care; Evidence-based guideline; Prematurity; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: parallel group (experimental-control)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single blinding (to mothers) was performed in this study. Care provider blinding was performed because the mothers did not know whether kangaroo care was carried out in accordance with a guide. In addition, because the premature babies in the study would not know which group they were in, participant blinding was performed.
  In order to prevent bias in the analysis phase of the data; Analysis was done by an independent statistician. After the statistical analysis was completed and the report of the research was prepared, it was explained how the intervention and control groups were coded. The intervention group was coded with '1' while the control group was coded with the number '2'.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Kangaroo care was applied for 65 minutes to premature infants by their mothers based on the kangaroo care guide.
  Interventions: Other: Kangaroo care based on kangaroo care guide
- Control Group (No Intervention): Kangaroo care was routinely administered by the nurse for 65 minutes without using a kangaroo care guide.

INTERVENTIONS:
Other: Kangaroo care based on kangaroo care guide — Under the supervision of the researcher, a kangaroo care practice was applied to premature babies by their mothers based on the kangaroo care guide. This practice took 65 minutes. In addition, before the application, the kangaroo application information was explained to the mothers through a brochure.
  Arms: Intervention Group

SUMMARY:
The aim of this study was to determine the effect of the use of clinical guidelines in kangaroo care (KB) practice on neonatal and maternal outcomes in premature infants.

The study was a single-blind, parallel group (experimental-control), randomized controlled experimental design with pretest-posttest design.

It was carried out in the neonatal intensive care unit of Selçuk University Faculty of Medicine Hospital in Konya province. Study data were collected from 40 premature newborns between September 2022 and November 2022. Premature infants in the intervention (n = 20) and control groups (n = 20) were determined by randomization method.

DETAILED DESCRIPTION:
Kangaroo care was applied to the intervention group with the Kangaroo Care Guide created by reviewing the current literature, and kangaroo care was applied to the control group with the standard kangaroo care method of the clinic. Data were collected using the Descriptive Information Form, Physiological Parameters Form, Neonatal Comfort Behavior Scale, Nurse-Parent Support Scale, Parental Satisfaction Scale and Kangaroo Care Guide/Checklist for Infants Without Respiratory Support.

Premature infants were followed up with skin-to-skin contact with their mothers in kangaroo care for 65 minutes. In the study, physiological parameters and Neonatal Comfort Behavior Scale scores of premature infants and Nurse-Parent Support Scale and Parental Satisfaction Scale scores of mothers were evaluated. Pearson Chi-Square Test, Yates Correction and Fisher's Exact Test were used to compare categorical data according to groups. Two Independent Sample t Test was used to compare normally distributed variables and Mann Whitney U Test was used to compare non-normally distributed variables. Statistical significance level was accepted as p˂0.05.

ELIGIBILITY:
Inclusion Criteria:

For premature infants;

* The baby is born before 36+6 weeks of gestation
* Stability of vital parameters at the time of application,
* Stable health status (cardiorespiratory stability, no congenital or chromosomal abnormalities, no history of intraventricular hemorrhage, no history of periventricular leukomalacia and NEC, no systemic and metabolic disorders),

For mothers;

* Willingness to participate in the research
* Being able to read and write Turkish

Exclusion Criteria:

For premature infants;

* Being connected to a mechanical ventilator
* Congenital or chromosomal abnormality
* Being with deprivation syndrome
* Having a history of intraventricular hemorrhage

For mothers; Not being willing to care for kangaroos

- Having a physical disability to care for kangaroos

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Physiological parameters of the premature infant:respiration rate | Change from baseline and 70 min
  The infant's is respiratory rate per minute.
Physiological parameters of the premature infant:peak heart rate | Change from baseline and 70 min
  The infant's is heart rate per minute. Philips IntelliVue MP40 device was used to monitor heart rete.
Physiological parameters of the premature infant: oxygen saturation | Change from baseline and 70 min
  Oxygen saturation measures the percentage of oxyhemoglobin (oxygen-bound hemoglobin) in the blood, and it is represented as arterial oxygen saturation (SaO2) and venous oxygen saturation (SvO2). Philips IntelliVue MP40 device was used to monitor %SpO2.
Physiological parameters of the premature infant: body temperature | Change from baseline and 70 min
  Shows body temperature.
Comfort Behavior scale scores of the premature infant | Change from baseline and 70 min
  Comfort Behavior scale was used. The Neonatal Comfort Behavior Scale (NEAS) is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. Each item in the scale is scored from 1 to 5. It is evaluated over the total score. The lowest score that can be obtained from the Newborn Comfort Behavior Scale (NEAS) is 6, and the highest score is 30.

SECONDARY OUTCOMES:
Parent Satisfaction points | baseline and 70 min
  Parental Satisfaction scale was used. This scale was developed to assess parents' satisfaction in NICU. EMPATHIC-30 scale, 1= definitely not; 6 = absolutely yes and consists of five sub-dimensions; information (5 items), care and treatment (8 items), organization (5 items), parent involvement (6 items) and the professional attitude of the staff (6 items). One point represents the lowest satisfaction, while 6 points represents the highest satisfaction.
Nurse Parent Support score | baseline and 70 min
  Nurse Parent Support scale was used. The scale consists of 21 items and four scales in five-point Likert type (1) "almost never", (2) "sometimes", (3) "sometimes", (4) "often" and (5) "always". consists of sub-scales; "Information and Communication Support" (9 items), "Emotional Support" (3 items), "Respect Support" (4 items), "Quality Care Giving" (5 items) (See Appendix E). The lowest score that can be obtained from the scale is 21, while the highest score is 105. A high score indicates that the support given by the nurse to the parent is high.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ayça Özkan, Principal Investigator — Konya Beyhekim Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya, Selcuklu
  - Selcuk University, Konya

IPD SHARING:
Plan to Share IPD: No